CLINICAL TRIAL: NCT01520623
Title: Role of Complement System in Human Allogeneic Haematopoietic Stem Cell Transplantation
Brief Title: Complement and Graft-versus-host Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Clinical haematology and BMT unit,Necker Hospital, Paris (Unknown); Clinical haematology and BMT unit,Saint Antoine Hospital, Paris (Unknown); Clinical haematology and BMT unit,Saint Louis Hospital,Paris (Unknown); European Georges Pompidou Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRC 08025
Record Dates: First submitted 2011-12-26; First posted 2012-01-30 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Allografted With Myeloablative Conditioning
Keywords: Allogeneic haematopoietic stem cell transplantation (HSCT); Myeloablative conditioning for an haematological malignancy; Graft-versus-host disease (GvHD); Activation of complement system; Gut GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allografted patients (Other): Allografted patients with myeloablative conditioning for an haematological malignancy. Patients will be followed for at least 12 months after transplantation and blood samples drawn before conditioning and once a week for 12 weeks after transplantation to analyze the serum concentration of Complement factors (C3, C4, B factor), Complement regulatory proteins (C1-inhibitor, I and H Factors) and analysis of the surface expression of Complement regulatory molecules such as CD46, CD55 and CD59 and the serum inflammatory cytokine levels
  Interventions: Other: Serum concentration /Serum inflammatory

INTERVENTIONS:
Other: Serum concentration /Serum inflammatory — Allografted patients with myeloablative conditioning for an haematological malignancy. Patients will be followed for at least 12 months after transplantation and blood samples drawn before conditioning and once a week for 12 weeks after transplantation to analyze the serum concentration of Complement factors (C3, C4, B factor), Complement regulatory proteins (C1-inhibitor, I and H Factors) and analysis of the surface expression of Complement regulatory molecules such as CD46, CD55 and CD59 and the serum inflammatory cytokine levels

SUMMARY:
Allogeneic haematopoietic stem cell transplantation (HSCT) often remains the only curative treatment for haematological malignancies. The anti-leukaemic effect of allogeneic HSCT, called the GvL (Graf-versus-Leukemia) effect, is often associated to the development of an immune response against healthy recipient cells leading to a graft-versus-host disease (GvHD) in 20 to 70% of allogeneic HSCT. Acute GvHD, that usually targets the skin, the gastrointestinal (GI) tract and the liver, is an important cause of morbidity and mortality after allogeneic HSCT, particularly in the case of GI GvHD. The main goal of the research in the field of allogeneic HSCT is to determine strategies that could decrease the risk of GvHD without affecting the GvL effect. According to GVHD experimental models, it is likely that GvL but not GvHD may occur in the absence of inflammatory signals induced by the transplant-associated conditioning. Based on this hypothesis, we have chosen to analyse the role of Complement system in patients who received allogeneic HSCT. Indeed, Complement system is a major actor of inflammation and in the generation of tissue destruction, both of which are involved in the physiopathology of GVHD. Furthermore, it might be a potential target of some available inhibitory drugs (purified C1-Inhibitor, anti-C5 antibodies) in a preventive or curative manner in such patients. Preliminary data obtained from 34 allografted patients in our institution suggest that Complement activation by the classical pathway is correlated to the occurrence of GI GVHD. The goal of our current project, in order to confirm these preliminary results in a larger series, is to explore Complement system activation in patients who received allogeneic HSCT in three Adult Hematology departments in Paris fot two years and to correlate the biological results to the clinical events occurring after HSCT.

DETAILED DESCRIPTION:
The study will be performed in allografted patients with myeloablative conditioning for an haematological malignancy from 3 adult transplant units.

Patients will be followed for at least12 months after transplantation and blood samples drawn before conditioning and once a week for 12 weeks after transplantation to analyze:

* serum concentration of Complement factors (C3, C4, B factor), Complement regulatory proteins (C1-inhibitor, I and H Factors) and analysis of the surface expression of Complement regulatory molecules such as CD46, CD55 and CD59.
* serum inflammatory cytokine levels

In addition, patients with clinical signs of gut GVHD will be explored by gastrointestinal endoscopy to perform gut biopsies. C5b9 deposure will be then analyzed by immunohistochemistry on GVHD lesions.

Activation of complement system will be defined by a decrease of complement factor levels of 50% and values under lower physiological limits. The clinical evolution and the inflammatory cytokine profile of patients with such an activation profile will be compared to that of those without complement activation.

A data base containing biological and clinical data will be established. Biological results will be correlated to post-transplant clinical events, in particular the occurrence of gut GVHD but also non relapse mortality and overall survival by adapted statistical tests (comparison of percentages by Chi-2 of Pearson, comparison of survival curves by logrank, multivariate analysis by logistic regression test or cox model).

The number of required patients will be established by comparison of the percentage of gut GVHD in the patients with or without complement activation. Based on our preliminary results, we hypothesize that 2/3 patients will not have complement activation among whose 20% will develop acute gut GVHD. We expect an increase of acute gut GVHD up to 60% of the patients with complement activation that would represent 1/3 of the cohort.

With a bilateral alpha risk of 5% and a power of 80%, the number of required patients is 23 in the activated group and 46 in the non activated group, thus a total of 69 patients.

ELIGIBILITY:
Inclusion Criteria:

* Allografted patients with myeloablative conditioning for an haematological malignancy
* Age > 18 years old and < 65 years.
* The patient must have access to social insurance according to local regulations.
* Patient must give a written informed consent (personally signed and dated) before completing any study related procedure

Exclusion Criteria:

* Age < 18 years old and > 65 years
* Patient with active infection HIV, HTLV1, Hepatite B ou C
* Uncontrolled infection(s), (i.e. documented bacterial, parasitical, or fungal infection).
* Patient with lupus
* Patient with transaminases > 5N, TP<30% with Facteur V < 30% before allogreffe
* Creatinine clearance < 50ml/min
* Absence of any psychological condition potentially hampering signing informed consent
* Patient refused to sign informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Activation of the complement system and the development of acute gut GvHD | 12 weeks
  Assessment of the activation of the complement system after human allogeneic stem cell transplantation and of its potential correlation with the development of acute gut GvHD

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall Survival at 3, 6, 9 , 12 and 24-month Post HCST
Overall survival without relapse | 2 Years
  Relapse

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Thérèse RUBIO, MD, PhD, Principal Investigator — Saint Antoine Hospital
Locations (3):
- France (3):
  - Saint Louis Hospital, Paris
  - Saint Antoine Hospital, Paris
  - Necker Hospital, Paris

REFERENCES:
- [Derived] Notarantonio AB, D'aveni-Piney M, Pagliuca S, Ashraf Y, Galimard JE, Xhaard A, Marcais A, Suarez F, Brissot E, Feugier P, Urien S, Bouazza N, Jacquelin S, Meatchi T, Bruneval P, Fremeaux-Bacchi V, Peffault De Latour R, Hermine O, Durey-Dragon MA, Rubio MT. Systemic complement activation influences outcomes after allogeneic hematopoietic cell transplantation: A prospective French multicenter trial. Am J Hematol. 2023 Oct;98(10):1559-1570. doi: 10.1002/ajh.27030. Epub 2023 Jul 22. PMID 37483161